CLINICAL TRIAL: NCT00555867
Title: A Randomised in Practice Evaluation of the Influence of Patient's Understanding of Her Disease and Therapy on Persistence and Compliance to Adjuvant Therapy for Post-menopausal Hormone Sensitive Early Breast Cancer
Brief Title: Patient's Anastrozole Compliance to Therapy Programme
Acronym: PACT
Status: Terminated | Type: Observational
Why Stopped: High drop-out rate leads to the conclusion: not enough data will be available to perform proper analyses of data collected after follow-up month 24 visit
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 1033GR/0002
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
Keywords: hormone-receptor positive primary breast cancer; compliance; Postmenopausal women
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance | interventions — Anastrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Standard routine care for breast cancer
  Interventions: Drug: Anastrozole
- 2: Standard + Intervention arm: standard routine care for breast cancer and additional information material via post
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — oral
  Other Names: Arimidex; ZD1033

SUMMARY:
Approximately 60 specialised clinics and 420 office based gynaecologists or oncologists will participate in this in practice evaluation program (NIS). The clinic and approximately 7 office based physicians will collaborate within their breast centre networks to conduct this program. A breast centre network should be able to recruit in this program approximately 80 patients (approximately 40 patients per year). It is planned to enroll approximately 4674 patients in this NIS (2337 patients per arm). The patient population will include postmenopausal women with hormone-receptor positive primary breast cancer scheduled for upfront adjuvant endocrine treatment with anastrozole according to the current standard medical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological confirmed primary diagnosis of early breast cancer
* Postmenopausal
* Hormone receptor positive

Exclusion Criteria:

* Patients with severe renal function disorders
* Patients with moderate or severe disorders of hepatic function
* Concomitant treatment with drugs known to affect sex hormonal status and tamoxifen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with hormone receptor positive primary breast cancer scheduled for upfront adjuvant endocrine treatment with anastrozole according to the current standard medical practice
Sampling Method: Probability Sample
Enrollment: 4923 (Actual)
Dates: Start 2006-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Compliance rate and persistence rate | until discontinuation of treatment

SECONDARY OUTCOMES:
Time to treatment discontinuation | date of last intake of anastrozole minus date of first prescription of anastrozole + 1
Demographics and other baseline characteristics as well as information regarding concomitant medication, quality of life | until treatment discontinuation
The percentage number of patients with disease free survival | after 12 months
Time of disease free survival | date of recurrence or progression of the tumor minus date of primary breast cancer surgery + 1

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Germany Medical Director, Study Director — AstraZeneca

REFERENCES:
- [Derived] Hadji P, Blettner M, Harbeck N, Jackisch C, Luck HJ, Windemuth-Kieselbach C, Zaun S, Kreienberg R. The Patient's Anastrozole Compliance to Therapy (PACT) Program: a randomized, in-practice study on the impact of a standardized information program on persistence and compliance to adjuvant endocrine therapy in postmenopausal women with early breast cancer. Ann Oncol. 2013 Jun;24(6):1505-12. doi: 10.1093/annonc/mds653. Epub 2013 Feb 1. PMID 23378537